CLINICAL TRIAL: NCT07010081
Title: Using Digital Health in a Postoperative Setting After Major Surgery: a Prospective Single-center Quantitative Survey Study
Brief Title: Using Digital Health in a Postoperative Setting After Major Surgery: Survey Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Professor, Dr, Jessa Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/047
Record Dates: First submitted 2025-05-27; First posted 2025-06-08 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Digital Health
Keywords: Remote monitoring; Major surgery
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surveys (Experimental): Conducting questionnaires during a follow-up consultation after major surgery
  Interventions: Procedure: Surveys

INTERVENTIONS:
Procedure: Surveys — Several questionnaires will be conducted once in-person to each patient after a follow-up consultation in the hospital after their major surgery

SUMMARY:
This study aims to explore patients' use of digital services for self-management of their health following major surgery at Jessa Hospital. Besides this, the study evaluates patients' ability to process and critically assess health information during recovery, their understanding of health concepts and risk factors, and their perception of data security and control over personal health information. Additionally, the study aims to examine patients' motivation to use digital services, their access to and trust in reliable digital health resources, and how well these services meet their individual needs. Furthermore, the study assesses the acceptability, appropriateness, and feasibility of using digital health tools in a post-operative setting, as well as evaluating the digital readiness of patients after surgery.

DETAILED DESCRIPTION:
Digital health technologies are transforming healthcare, offering new ways to improve patient outcomes and enhance efficiency. Remote clinical monitoring (RCM), which uses digital technologies such as wearable devices and mobile apps to monitor patients outside of the traditional healthcare settings such as a hospital, holds significant potential for supporting post-operative care, especially in the context of faster hospital discharge after major surgery. Major surgery involves procedures on organ systems, such as cancer resections, organ transplants, and lung or abdominal surgeries. However, despite their promise, the successful implementation of these technologies into clinical practice requires a thorough understanding of the perspectives of the end user, being the patient. Patients' comfort, engagement, and perceptions about digital health solutions, such as self-management tools and remote monitoring pathways, are essential to ensuring these technologies are both effective and widely accepted.

ELIGIBILITY:
Inclusion Criteria:

* Surgical patients

  * >18 years old, Undergone major surgery at Jessa Hospital Hasselt

Exclusion Criteria:

* Unable to provide informed consent or request to not participate in the study
* Cognitively incapable of understanding the study
* No understanding of the Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Patients' understanding of comfort and engagement with using digital services for self- management of their disease | During a follow-up consultation within one year after major surgery
  The patients' understanding of comfort and engagement with using digital services for self- management of their disease after major surgery will be evaluated using scale 4 of the eHLQ.

SECONDARY OUTCOMES:
Ability of patients to use technology to process and critically evaluate health information | During a follow-up consultation within one year after major surgery
  The ability of patients to use technology to process and critically evaluate health information during postoperative recovery will be evaluated using scale 1 of the eHLQ.
Patients' understanding of health concepts, their health status, and risk factors | During a follow-up consultation within one year after major surgery
  Scale 2 of the eHLQ will assess patients' understanding of health concepts, their health status, and risk factors during their recovery period.
Patients' perception of data security and control over personal health data | During a follow-up consultation within one year after major surgery
  To assess patients' perception of data security and control over personal health data in digital services, scale 4 of the eHLQ will be used.
Patients' motivation to use digital services for managing postoperative health | During a follow-up consultation within one year after major surgery
  Scale 5 of the eHLQ is used to examine patients' motivation to use digital services for managing their postoperative health.
Patients' access to and trust in reliable digital health services | During a follow-up consultation within one year after major surgery
  The sixth scale of the eHLQ will evaluate patients' access to and trust in reliable digital health services during recovery.
The extent to which digital health services meet patients' individual needs and preferences | During a follow-up consultation within one year after major surgery
  To assess how well digital health services meet patients' individual needs and preferences during recovery, scale 7 of the eHLQ will be used.
Acceptability, appropriateness, and feasibility of using digital health by means of implementation outcome measures AIM, IAM, and FIM | During a follow-up consultation within one year after major surgery
  To evaluate the acceptability, appropriateness, and feasibility of using digital health in a postoperative setting after major surgery, the AIM, IAM, and FIM, respectively, will be used.
Digital readiness | During a follow-up consultation within one year after major surgery
  The DHRQ will be used to assess digital readiness of patients that underwent major surgery.
External validation of the digital health readiness questionnaire | During a follow-up consultation within one year after major surgery
  The DHRQ will be externally validated against the extensively validated eHLQ.

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium